CLINICAL TRIAL: NCT00532415
Title: Clinical Evaluation of the Safety and Efficacy of Triamcinolone Acetonide Suspension for Visualization During Vitrectomy Surgery
Brief Title: Safety and Efficacy of Vitreous Delineating Agent During Vitrectomy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: C-05-62
Record Dates: First submitted 2007-09-19; First posted 2007-09-20 (Estimated); Last update posted 2012-04-05 (Estimated); Status verified 2012-04

CONDITIONS: Vitrectomy
Keywords: Vitrectomy; Visualization

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (1):
- Triamcinolone (Experimental): Approximately 1-4 mg (0.025-0.1 cc) as needed for visualization during pars plana vitrectomy with or without membrane removal.
  Interventions: Drug: Triamcinolone Acetonide Injectable Suspension

INTERVENTIONS:
Drug: Triamcinolone Acetonide Injectable Suspension — Approximately 1-4 mg (0.025-0.1 cc) as needed for visualization during pars plana vitrectomy with or without membrane removal.

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of triamcinolone acetonide suspension when used for visualization of structures in the back of the eye during eye surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients planning to undergo pars plana vitrectomy with good vision in the non-surgery eye.
* Other protocol-defined inclusion criteria may apply.

Exclusion Criteria:

* Patients under 18.
* Patients with previous vitrectomy, elevated intraocular pressure (IOP) and/or history of ocular inflammatory disease.
* Other protocol-defined exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2007-09; Primary Completion 2007-09 (Actual); Study Completion 2007-09 (Actual)

PRIMARY OUTCOMES:
Change in Mean Visualization Score at Post-Instillation from Pre-Instillation | Day 0
  A video image of the posterior segment structures of the eye was taken before instillation of the test product and after. An independent masked reader evaluated the images and graded the degree of visualization on a 5-point scale ranging from 1 to 4 and anchored at the ends by "Not Visible (0)" and "Clearly Delineated (4)." The mean difference was calculated, and a higher number indicated increased visibility.